CLINICAL TRIAL: NCT02958930
Title: An Open-Label Study to Evaluate the Safety and Efficacy of Transcranial Electromagnetic Treatment (TEMT) for the Treatment of Alzheimer's Disease
Brief Title: Safety and Efficacy of Transcranial Electromagnetic Treatment Against Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroEM Therapeutics, Inc. (Industry)
Collaborators: Byrd Alzheimer's Institute, University of South Florida (Unknown); University Diagnostic Institute, Tampa (Unknown); Invicro, Boston (Unknown); Left Coast Engineering, Escondido (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeuroEM-001; EM 1000-1 (Other: TBA)
Record Dates: First submitted 2016-11-01; First posted 2016-11-08 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Alzheimer Disease; Alzheimer Disease, Late Onset
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TEMT Treatment (Experimental): Patients in this arm will receive Transcranial Electromagnetic Treatment (TEMT) twice daily for a two-month treatment period utilizing the MemorEM 1000 head device.
  Interventions: Device: MemorEM 1000

INTERVENTIONS:
Device: MemorEM 1000 — The MemorEM 1000 device is self-contained and has been designed for in-home daily electromagnetic treatment in the radiofrequency range, allowing for complete mobility and comfort in performing daily activities during treatment. The device has a custom control panel that is powered by a rechargeable battery. This control panel/battery box is worn on the upper arm and wired to specialized antennas in the head cap worn by the subject. The device provides global RF treatment to the entire forebrain, including deep brain areas. For each of the 60 days of in-home treatment, two one-hour treatment will be given (early morning and late afternoon). Each treatment will be administered by the patient's caregiver, who will position the device on the patient's head and monitor treatment.

SUMMARY:
The purpose of this study is to determine the safety and initial efficacy of Transcranial Electromagnetic Treatment (TEMT) in patients with mild/moderate Alzheimer's Disease. Throughout a 2-month treatment period, patients will be evaluated for cognitive performance, brain energy utilization, functional brain imaging, and blood/cerebrospinal fluid (CSF) markers for Alzheimer's Disease. Since all patients will receive TEMT, each patient's baseline measurements will serve as their own control for any treatment effects.

DETAILED DESCRIPTION:
There is currently no effective therapeutic to stabilize or reverse the cognitive impairment of Alzheimer's Disease (AD) and related dementias. Clinical trials with drugs have been unsuccessful because the wrong therapeutic target/species were selected, because drugs have great difficulty traversing the blood-brain barrier and getting into neurons, and/or because drugs largely have only a single mechanism of action. Since ever-increasing experimental evidence indicates that the toxic forms of both beta-amyloid and tau are the soluble "oligomeric" species of these two proteins, therapeutics to disaggregate these oligomers within neurons represent perhaps the best chance for attaining cognitive benefit in AD patients.

Pre-clinical studies performed by the Sponsor and his collaborators have demonstrated that AD transgenic mice treated daily with electromagnetic waves in the radiofrequency (RF) range are protected from cognitive impairment or show a reversal of pre-existing cognitive impairment. These cognitive benefits appear to be due primarily to two complimentary mechanisms: 1) disaggregation of toxic protein oligomers within neurons, and 2) mitochondrial enhancement to increase energy metabolism. Moreover, no deleterious effects of treatment over many months have been observed in these pre-clinical studies.

In order to provide similar treatment to mild/moderate Alzheimer's patients clinically, NeuroEM Therapeutics has developed a unique head device that provides electromagnetic (RF) treatment to the entire human forebrain at levels similar to those that provided cognitive benefits in pre-clinical studies. Using the MemorEM 1000 head device in the present Phase I trial, AD patients receive twice daily 1-hour treatments in-home, as administered by their caregiver. The device allows for the patient to have complete mobility for moving throughout their home.

A comprehensive array of markers will be analyzed both during and following the 2-month treatment period, with baseline (pre-treatment) values serving as controls. Cognitive safety and efficacy will be evaluated using a variety of cognitive assessments including ADAS-cog (Primary), and secondary cognitive measures including ADCS-ADL, Rey AVLT, Trails A & B, Digit span, and clock draw tasks. Treatment effects on brain energy metabolism will be determine by FDG-PET scans, while treatment effects on brain functional connectivity will be determined through both resting state MRI and Diffusion Tensor Imaging. Also being assessed are the effects of treatment on various beta-amyloid and tau protein species (e.g., monomers, oligomers) in both blood and CSF. Safety of the treatment will be monitored by regular Adverse Events Assessment, physiologic monitoring, and patient daily diaries maintained by the caregiver.

Expected Results: The investigators expect that 2-months of daily electromagnetic (RF) treatment will not present any significant side effects or safety issues. The investigators further expect that cognitive measures will be stable and/or improve by the end of treatment. In addition, the investigators anticipate that brain functional connectivity may be improved and that enhanced brain metabolism (FDG-PET) will occur. Changes in blood/CSF levels of various beta-amyloid and tau species are also anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mild or moderate stage of Alzheimer's Disease, according to the National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
* MMSE score 16 to 26
* Physical clearance for study participation as evaluated by the clinician.
* Caregiver (spouse, family member, etc.) who agrees to and is capable of taking care and being responsible for the participation of the patient in the study (keeping a diary of health measures they collect on the patient at home, logging the patient's condition daily, and assuming responsibility for administering daily in-home treatment). Caregiver to have non-impaired mental abilities and normal motor skills, as determined by the investigators at screening. The definition of caregivers for this study is adults providing unpaid care to relatives or friends to help them take care of themselves in such activities as managing finances, shopping, preparing meals, and going to doctor appointments.
* Agreement to participate in approximately 10 weeks during the study.
* Normal to near-normal vision and hearing with correction as needed (e.g. corrective lenses, hearing aid).
* Fluent in English
* Minimum of 8th grade education
* Head circumference between 53 - 58 cm (to minimize variability in head antenna locations)
* If medicated for AD, then use of cholinesterase inhibitors and/or memantine for at least 3 months, on stable dose for at least 60 days prior to screening, and maintenance on that dose for the period of this study.
* All other non-AD medications must be stable for a period of 4 weeks prior to screening

Exclusion Criteria:

* CDR Global Score of 0, 0.5 or 3
* Severe agitation
* Mental retardation
* Unstable medical condition
* Use of benzodiazepines or barbiturates 2 weeks prior to screening
* Participation in a clinical trial with any investigational agent within 6 months prior to study enrollment and no history of immunotherapy research participation
* History of Epileptic Seizures or Epilepsy
* Patients with major depression (not controlled with medication), bipolar disorder or psychotic disorders or any other neurological or psychiatric condition (whether now or in the past). The investigator will obtain this information from available patient medical records, history provided by the patient and caregiver, interview, and neurological exam.
* Alcoholism or drug addiction as defined by DSM-IV within last 5 years (addicted more than one year and or in remission less than 3 years) or severe sleep deprivation
* Patients with metal implants in the head, (i.e. cochlear implants, implanted brain stimulators, aneurysm clips) with the exception of metal implants in mouth
* Patients with vitamin B12 deficiency, abnormal thyroid function, or personal history of either any clinically defined medical disorder or any clinically defined neurological/psychiatric disorder (other than AD), including (but not limited to):, stroke, brain lesions, , cerebrovascular condition, other neurodegenerative disease, significant head trauma (loss of consciousness greater than half an hour, or related anterograde amnesia), multiple sclerosis; or personal history of previous neurosurgery or brain radiation
* Patients with any signs or symptoms of increased intracranial pressure, as determined in a neurological exam.
* Patients with demonstrated brain micro-hemorrhages at screening
* Patients with a score of 4 or higher on the Hachinski Test
* Patients with a score of 2 or less on the Global Deterioration Scale
* Patients with hypertension that is unresponsive to anti-hypertensive medications
* Patients with a history of migraine headaches occurring more than once a month
* Patients with a history of cancer within the last 3 years
* Patients chronically taking anticoagulants or anti-platelets (at discretion of Principal Investigator)
* Pregnant women and women who have the ability to become pregnant
* Patients with compressed hair thickness of more than 5mm (which could increase distance between head antennas and the scalp).
* Cardiac pacemakers
* Implanted medication pumps
* Intracardiac lines
* Significant heart disease

Min Age: 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
ADAS-Cog | Change from baseline ADAS-Cog at 2 months
  ADAS-Cog is the standard/benchmark test of cognitive performance evaluated in Alzheimer's-related clinical trials.

SECONDARY OUTCOMES:
FDG-PET | Change from baseline FDG-PET at 2 months
  FDG-PET scanning is used to determine brain energy metabolism/utilization
Resting state fMRI | Change from baseline rsfMRI at 2 months
  rsfMRI is an MRI scan used to evaluate brain functional connectivity
Diffusion Tensor Imaging (DTI) | Change from baseline DTI at 2 months
  DTI is an MRI scan used to evaluate brain functional connectivity
Susceptibility-Weighted Imaging (SWI) | Change from Baseline SWI at 2 months
  SWI is an MRI scan used to determine any brain microhemorrhages or tumors
Blood and CSF beta-amyloid levels | Change from Baseline beta-amyloid levels at 2 months
  Blood and CSF will be analyzed for the toxic protein beta-amyloid
Blood and CSF tau levels | Change from Baseline tau levels at 2 months
  Blood and CSF will be analyzed for the toxic protein tau
Blood and CSF markers of immune function | Change from Baseline pro- and anti-inflammatory cytokine levels at 2 months
  Blood and CSF will be analyzed for pro- and anti-inflammatory cytokines (same measure units)
Blood and CSF markers of oxidative stress | Change from Baseline oxidative stress levels at 2 months
  Blood and CSF will be analyzed for oxidative markers (same measure units)
Adverse Event Assessment | Change from Baseline Adverse Event Assessment at 2 months
  AEA will be the primary safety outcome measure
ADCS-ADL score | Change from Baseline ADCS-ADL score at 2 months
  This is a secondary cognitive outcome to assess effects of treatment on cognition.
MMSE score | Change from Baseline MMSE score at 2 months
  This is a secondary cognitive outcome to assess effects of treatment on cognition.
Global Deterioration score | Change from Baseline Global Deterioration score at 2 months
  This is a secondary cognitive outcome to assess effects of treatment on cognition.
Hachinski score | Change from Baseline Hachinski score at 2 months
  This is a secondary cognitive outcome to assess effects of treatment on cognition.
Rey AVLT score | Change from Baseline Rey AVLT score at 2 months
  This is a secondary cognitive outcome to assess effects of treatment on cognition.
Trails A & B score | Change from Baseline Trails A & B scores at 2 months
  This is a secondary cognitive outcome to assess effects of treatment on cognition.
Digit span score | Change from Baseline Digit span score at 2 months
  This is a secondary cognitive outcome to assess effects of treatment on cognition.
Clock draw score | Change from Baseline Clock draw score at 2 months
  This is a secondary cognitive outcome to assess effects of treatment on cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Smith, MD, Principal Investigator — Byrd Alzheimer's Institute, University of South Florida
Locations (1):
- Byrd Alzheimer's Institute, University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
It is not anticipated that IPD will be shared with other researchers

REFERENCES:
- [Background] Arendash GW. Review of the Evidence that Transcranial Electromagnetic Treatment will be a Safe and Effective Therapeutic Against Alzheimer's Disease. J Alzheimers Dis. 2016 May 30;53(3):753-71. doi: 10.3233/JAD-160165. PMID 27258417
- [Background] Arendash GW. Transcranial electromagnetic treatment against Alzheimer's disease: why it has the potential to trump Alzheimer's disease drug development. J Alzheimers Dis. 2012;32(2):243-66. doi: 10.3233/JAD-2012-120943. PMID 22810103
- [Background] Arendash GW, Mori T, Dorsey M, Gonzalez R, Tajiri N, Borlongan C. Electromagnetic treatment to old Alzheimer's mice reverses beta-amyloid deposition, modifies cerebral blood flow, and provides selected cognitive benefit. PLoS One. 2012;7(4):e35751. doi: 10.1371/journal.pone.0035751. Epub 2012 Apr 25. PMID 22558216
- [Background] Dragicevic N, Bradshaw PC, Mamcarz M, Lin X, Wang L, Cao C, Arendash GW. Long-term electromagnetic field treatment enhances brain mitochondrial function of both Alzheimer's transgenic mice and normal mice: a mechanism for electromagnetic field-induced cognitive benefit? Neuroscience. 2011 Jun 30;185:135-49. doi: 10.1016/j.neuroscience.2011.04.012. Epub 2011 Apr 13. PMID 21514369
- [Background] Arendash GW, Sanchez-Ramos J, Mori T, Mamcarz M, Lin X, Runfeldt M, Wang L, Zhang G, Sava V, Tan J, Cao C. Electromagnetic field treatment protects against and reverses cognitive impairment in Alzheimer's disease mice. J Alzheimers Dis. 2010;19(1):191-210. doi: 10.3233/JAD-2010-1228. PMID 20061638
- [Background] Mori T, Arendash GW. Electromagnetic field treatment enhances neuronal activity: Linkage to cognitive benefit and therapeutic implications for Alzheimer's Disease. J Alzheimer's Dis and Parkinsonism 2011: Vol. 1:102, http://dx.doi.org/10.4172/2161-0460.1000102.
- [Derived] Cao C, Abulaban H, Baranowski R, Wang Y, Bai Y, Lin X, Shen N, Zhang X, Arendash GW. Transcranial Electromagnetic Treatment "Rebalances" Blood and Brain Cytokine Levels in Alzheimer's Patients: A New Mechanism for Reversal of Their Cognitive Impairment. Front Aging Neurosci. 2022 May 2;14:829049. doi: 10.3389/fnagi.2022.829049. eCollection 2022. PMID 35585867
- See also: Website provides additional information regarding this technology — http://www.neuroem.com